CLINICAL TRIAL: NCT06632457
Title: A Phase III Double-blind, Randomised, Placebo-controlled Trial to Evaluate Liver-related Clinical Outcomes and Safety of Once Weekly Injected Survodutide in Participants With Compensated Non-alcoholic Steatohepatitis/Metabolic Dysfunction Associated Steatohepatitis (NASH/MASH) Cirrhosis
Brief Title: LIVERAGE™ - Cirrhosis: A Study to Test Whether Survodutide Helps People With a Liver Disease Called NASH/MASH Who Have Cirrhosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1404-0064; 2024-513741-36-00 (Registry Identifier: CTIS (EU)); U1111-1307-0227 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction Associated Steatohepatitis
MeSH Terms: interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Survodutide (Experimental)
  Interventions: Drug: Survodutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching survodutide

INTERVENTIONS:
Drug: Survodutide — Subcutaneous injection
  Other Names: BI 456906
  Arms: Survodutide
Drug: Placebo matching survodutide — Subcutaneous injection
  Arms: Placebo

SUMMARY:
This study is open to adults who are at least 18 years old and have:

* A confirmed liver disease called non-alcoholic steatohepatitis (NASH) or
* A confirmed liver disease called metabolic-associated steatohepatitis (MASH)
* BMI of 27 kg/m2 or more or
* 25 kg/m2 or more if the participant is Asian.

People with a history of other chronic liver diseases or high alcohol intake cannot take part in this study. The purpose of this study is to find out whether a medicine called survodutide helps people with NASH or MASH improve their liver function.

Participants are put into 2 groups randomly, which means by chance. 1 group gets survodutide and 1 group gets placebo. Placebo looks like survodutide but does not contain any medicine. Each participant has twice the chance of getting survodutide. Participants and doctors do not know who is in which group. Participants inject survodutide or placebo under their skin once a week. All participants regularly receive counselling to make changes to their diet and to exercise regularly.

Participants are in the study for up to 4 and a half years. During this time, they visit the study site or have a remote visit by video call every 2, 4 or 6 weeks for about a 1 year and 5 months. After this time participants visit the trial site or have a remote visit every 3 months until the end of the study.

The doctors check participants' health and take note of any unwanted effects. The participants' body weight is regularly measured. At some visits the liver parameters are measured using different imaging methods. The participants also fill in questionnaires about their symptoms. The results are compared between the groups to see whether the treatment works.

ELIGIBILITY:
Inclusion criteria:

1. Male or female adults ≥18 years of age at the time of screening, and at least the legal age of consent in countries where it is >18 years
2. Body mass index (BMI) ≥27 kg/m2(≥25 kg/m2 for Asian trial participants)
3. Compensated metabolic dysfunction-associated steatohepatitis (MASH) cirrhosis.
4. Magnetic resonance imaging proton density fat fraction (MRI-PDFF) fat fraction ≥5% or FibroScan® with controlled attenuation parameter (CAP) ≥288 dB/m, obtained during the screening period or a historic MRI-PDFF ≤12 weeks prior to randomisation (except for patients with 'cryptogenic cirrhosis' where MRI-PDFF <5% or FibroScan® with CAP <288 dB/m is allowed). This inclusion criterion does not apply for participants with a recent (≤12 months prior to randomisation) liver biopsy showing steatosis/steatohepatitis.
5. Further inclusion criteria apply.

Exclusion criteria:

1. Current or history (<5 years) of significant alcohol consumption, defined as an average of >140 g/week in female patients and >210 g/week in male patients, for a period of >3 consecutive months, or an inability to reliably quantify alcohol consumption based upon judgment of the investigator.
2. Model of end-stage liver Disease (MELD) score >12 due to liver disease
3. History or current (i.e. at screening) hepatic decompensation event of any of the following but not limited to:

   * Portal hypertension-related upper gastrointestinal (GI) bleeding
   * Ascites
   * Hepatic encephalopathy (HE) ≥Grade 1 according to the West Haven criteria
4. Any of the following lab test result at screening

   * Albumin below <3.5 g/dL (<35.0 g/L)
   * International normalised ratio (INR) >1.3 unless due to therapeutic anticoagulants
   * Total bilirubin (TBL) >1.2x upper limit of normal (ULN) NOTE: Trial participants with Gilbert Syndrome are eligible with a TBL >1.2x ULN if reticulocyte count is within normal limits, haemoglobin is within normal limits unless due to chronic anaemia and unrelated to haemolysis, and direct bilirubin is <20% of TBL.
   * Alkaline phosphatase >1.5x ULN
   * PLT <100,000/µL (<100 GI/L)
5. History or evidence of other chronic liver diseases, such as primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis or overlap syndrome, Wilson's disease, alpha-1-antitrypsin deficiency, or genetic haemochromatosis
6. Hepatitis B positive (defined as positive hepatitis B surface antigen (HBsAg)) or history of chronic HBV infection
7. Hepatitis C positive (defined as positive hepatitis C virus (HCV) antibody and a positive HCV ribonucleic acid (RNA))
8. Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >5x ULN
9. Evidence of alcoholic liver disease, or drug-induced liver disease, as defined on the basis of typical exposure and history
10. History of liver transplantation or listed for liver transplantation
11. History of transjugular intrahepatic portosystemic shunt (TIPS) or other radiological/surgical procedure for portal hypertension treatment
12. Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1590 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2029-06-05 (Estimated); Study Completion 2029-06-05 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of any component of the composite clinical endpoint (at EoS) consisting of: all-cause mortality, liver transplant, hepatic decompensation events, worsening of MELD score to ≥15 and progression to CSPH | up to 4.5 years.
  MELD = model of end-stage liver disease CSPH = Clinically significant portal hypertension

SECONDARY OUTCOMES:
Key secondary endpoint: Absolute change from baseline in enhanced liver fibrosis (ELF) score | At baseline and at Week 76.
Key secondary endpoint: Percentage change from baseline in body weight | At baseline and at Week 76.
Key secondary endpoint: Absolute change from baseline in glycosylated haemoglobin A1c (HbA1c) (%) in participants with type 2 diabetes mellitus (T2DM) at baseline | At baseline and at Week 76.
Key secondary endpoint: Absolute change from baseline in liver stiffness (kPa) in FibroScan® vibration-controlled transient elastography (VCTE) | At baseline and at Week 76.
Percentage change from baseline in liver stiffness in FibroScan® VCTE | At baseline and at Week 76.
Time to first occurrence of progression to CSPH | up to 4.5 years.
Time to first occurrence of any of the hepatic decompensation events (ascites, HE, or portal hypertension-related upper GI bleeding), or worsening of MELD score to ≥15 | up to 4.5 years.
Occurrence of all-cause hospitalisation (first and recurrent) | up to 4.5 years.
Time to first occurrence of any of the adjudicated components of the composite endpoint 5-point major adverse cardiac event (5P-MACE) | up to 4.5 years.
Absolute changes from baseline in lipids (mg/dL) | At baseline and at Week 76.
Absolute change from baseline in aspartate aminotransferase (AST) (U/L) | At baseline and at Week 76.
Absolute change from baseline in alanine aminotransferase (ALT) (U/L) | At baseline and at Week 76.
Absolute change from baseline in liver stiffness (kPa) assessed by magnetic resonance elastography (MRE) | At baseline and at Week 76.

CONTACTS AND LOCATIONS:
Locations (424):
- United States (121):
  - The Institute for Liver Health II DBA Arizona Clinical Trials, Peoria, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Velocity Clinical Research-Chula Vista, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - ARK Clinical Research, Fountain Valley, California
  - Velocity Clinical Research-Huntington Park, Huntington Park, California
  - 310 Clinical Research, Inglewood, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Om Research, LLC, Lancaster, California
  - Catalina Research Institute, LLC - Montclair, Montclair, California
  - Clinnova Research Solutions, Orange, California
  - Fomat Medical Research, Oxnard, California
  - Cadena Care Institute, Llc, Poway, California
  - Ficramed Research Institute, Poway, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Metro Clinical Trials, San Bernardino, California
  - Acclaim Clinical Research, San Diego, California
  - Future Innovative Treatments, Colorado Springs, Colorado
  - South Denver Gastroenterology PC, Englewood, Colorado
  - Connecticut Gastroenterology Clinical Research Foundation, Bristol, Connecticut
  - Synergy Healthcare, Brandon, Florida
  - Access research Institute, Brooksville, Florida
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - Top Medical Research, Inc, Cutler Bay, Florida
  - Covenant Metabolic Specialists, LLC - Fort Myers, Fort Myers, Florida
  - Neoclinical Research, Hialeah, Florida
  - Evolution Clinical Trials, Hialeah Gardens, Florida
  - Global Research Associates, Homestead, Florida
  - Lake Center for Clinical Research, Lady Lake, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Optimus U Corporation-Miami-69452, Miami, Florida
  - Schiff Center Liver Diseases, Miami, Florida
  - BioMed Research & Medical Center, Miami, Florida
  - MplusM - Century Research, Miami, Florida
  - ECIR Miami Holdings LLC dba IMIC, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Charter Research, Orlando, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Endoscopic Research, Inc, Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - MplusM - Best Choice Medical and Research Service, Pembroke Pines, Florida
  - Covenant Metabolic Specialist, LLC - Riverview, Riverview, Florida
  - Global Clinical Professionals, St. Petersburg, Florida
  - Synergy Healthcare, St. Petersburg, Florida
  - International Center for Research, Tampa, Florida
  - Charter Research, The Villages, Florida
  - Covenant Metabolic Specialists, LLC - University Park, University Park, Florida
  - Conquest Research, Winter Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - EmVenio Research-Atlanta-69582, Riverdale, Georgia
  - ASHA Clinical Research - Munster, LLC, Hammond, Indiana
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Tandem Clinical Research, Marrero, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Clinical Research Institute of Michigan, LLC, Clinton Township, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - MNGI Digestive Health, PA, Minneapolis, Minnesota
  - ObjectiveHealth-GI Associates Research, Columbia, Missouri
  - Kansas City Gastroenterology & Hepatology Physicians Group, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jubilee Clinical Research, Inc, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - IMA Clinical Research-Warren-69742, Warren Township, New Jersey
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Basil Clinical, Laurelton, New York
  - University of Rochester Medical Center, Rochester, New York
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Carolina Researche, Greenville, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - ObjectiveHealth-DSI Research, Springboro, Ohio
  - Northshore Gastroenterology Research, Westlake, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - US Digestive Health, Flourtown, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - US Digestive Health, Lancaster, Pennsylvania
  - US Digestive Health, Wyomissing, Pennsylvania
  - ObjectiveHealth-Columbia Digestive Health Research, Columbia, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Premier Medical Group, Clarksville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - IMA Clinical Research Austin, Austin, Texas
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Velocity Clinical Research, Austin, Austin, Texas
  - Pinnacle Clinical Research, LLC, Bellaire, Texas
  - South Texas Research Institute-Brownsville-68426, Brownsville, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Soma Clinical Trials, Denison, Texas
  - EmVenio Research Center at Prime Healthcare, Garden City, Texas
  - DHAT Reseach Institute, Garland, Texas
  - Pinnacle Clinical Research, LLC, Georgetown, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Research Physicians Network, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - GI Alliance, Mansfield, Texas
  - Biopharma Informatic LLC, McAllen, Texas
  - Centex Studies, Inc., McAllen, Texas
  - North Texas Research Institute - Dallas, Mesquite, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - HASresearch, San Antonio, Texas
  - Velocity Clinical Research, Waco, Waco, Texas
  - Objective Health-Digestive Research of Central Texas, Waco, Texas
  - ObjectiveHealth-Digestive Health Research of North Texas, Wichita Falls, Texas
  - GI Select Health Research LLC, Richmond, Virginia
  - Velocity Clinical Research-Seattle-69881, Seattle, Washington
  - Velocity Clinical Research-Spokane-69716, Spokane, Washington
- Argentina (9):
  - CIPREC, Buenos Aires
  - IDIM - Instituto de Diagnostico e Investigaciones Metabolicas, Buenos Aires
  - Buenos Aires Macula S.A., Buenos Aires
  - Glenny Corp - Centro Médico Saavedra, Buenos Aires
  - Centro de Investigaciones Metabolicas (CINME)-C.A.B.A-61553, C.a.b.a
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - Hospital Universitario Austral, Pilar
  - DIM Clinica Privada, Ramos Mejía
  - Hospital El Cruce, San Juan Bautista
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (5):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Ordensklinikum Linz GmbH, Linz
  - AKH - Medical University of Vienna, Vienna
  - Hospital Hietzing, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (5):
  - Hospital Universitário João de Barros Barreto, Belém
  - Hospital das Clinicas da Faculdade de Medicina da USP, Cerqueira César
  - Hospitalar Moinhos de Vento, Porto Alegre
  - Universidade Federal do Rio Grande do Sul, Porto Alegre
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
- Bulgaria (7):
  - MHAT Sv. Ivan Rilski EOOD, Gorna Oryahovitsa
  - Multi-profile Hospital For Active Treatment-Uni Hospital Ltd., Panagyurishte
  - Acibadem City Clinic Tokuda University Hospital EAD, Sofia
  - Diagnostic Consultative Center Alexandrovska, Sofia
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski EAD, Sofia
  - Medical Military Academy MHAT Sofia, Sofia
  - Medical Center New Rehabilitation Center EOOD, Stara Zagora
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Viable Clinical Research, Bridgewater, Nova Scotia
  - Toronto Liver Centre, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Centre de Médecine Métabolique de Lanaudière, Terrebonne, Quebec
  - Diex Recherche Québec, Québec
- Chile (3):
  - Edificio Fleming, La Serena
  - Centro de Investigaciones Médicas UC, Santiago
  - Centro de Investigaciones Clinicas Viña del Mar, Viña del Mar
- China (46):
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Provincial People's Hospital, Changsha
  - Changzhou Third People's Hospital, Changzhou Shi
  - West China Hospital, Sichuan University, Chengdu
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangzhou Eighth People's Hospital,Guangzhou Medical University, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - NanFang Hosptial, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - The First hospital of Jiaxing, Jiaxing
  - First People's hospital of Yunann Province, Kunming
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - The Second Hospital of Nanjing, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - Ningbo Second Hospital, Ningbo
  - General Hospital of Ningxia Medical University, Ningxia
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Renji Hospital Shanghai Jiaotong Univesrity School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Renmin Hospital of Wuhan University, Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - The Fifth People's Hospital of Suzhou, Suzhou
  - Tianjin Third Central Hospital, Tianjin
  - Tianjin Second People's Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Sixth People's Hospital of Zhengzhou, Zhengzhou
  - The Third People's Hospital of Zhenjiang, Zhenjiang
- Czechia (3):
  - Krajska nemocnice Liberec a.s., Liberec
  - Research Site s.r.o., Pilsen
  - General Faculty Hospital, Prague, Prague
- France (14):
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire D'Angers, Angers
  - Hôpital Beaujon, Clichy
  - HOP Dijon-Bourgogne, Côte-d'Or
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier De Versailles, Le Chesnay
  - Hopital De La Croix-Rousse, Lyon
  - Hôpital de l'Archet, Nice
  - Hôpital Claude Huriez, Nord-Pas-de-Calais
  - Hopitaux Universitaires Pitié-Salpétrière, Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire De Bordeaux, Passec
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
- Georgia (2):
  - Ltd "Health", Batumi
  - ISR-GEO Med Res Clin Healthycore, Tbilisi
- Germany (14):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Bochum
  - Universitätsklinikum Köln (AöR), Cologne
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universität des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Universitätsklinikum Münster, Münster
  - St. Josefs-Hospital Wiesbaden, Wiesbaden
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Hungary (2):
  - Obudai Egeszegugyi Centrum, Budapest
  - Semmelweis Egyetem Sebeszeti, Transzplantacios es Gasztroenterologiai Klinika, Budapest
- India (14):
  - Aryav Superspeciality Hospital, Ahemdabad
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Osmania Medical College & Hospital, Hyderabad, Afzalgunj
  - SR Kalla Memorial Hospital, Jaipur
  - ManglamPlus Medicity Hospital, Jaipur
  - G S V M, Kanpur, Kanpur
  - Atharva Multispecialty Hospital and research Centre, Lucknow
  - Midas Multispeciality Hospital Pvt Ltd, Nagpur
  - Insitute of Liver and Billiary Sciences, New Delhi
  - Pandit Bhagwat Dayal Sharma Post Graduate Institute of Medical Sciences, Rohtak
  - Yashoda Hospitals - Secunderabad, Secunderabad
  - Surat Institute of Digestive Sciences, Surat
  - BAPS Pramukh Swami Hospital, Surat
  - Gujarat Gastro and Vascular Hospital, Surat
- Italy (8):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Università degli Studi di Genova, Modena
  - Policlinico "Paolo Giaccone", Palermo
  - Fondazione Policlinico Universitario Campus Bio-medico, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Universita Degli Studi di Torino, Torino
- Japan (49):
  - The University of Tokyo Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Ehime University Hospital, Ehime, Toon
  - Fukuiken Saiseikai Hospital, Fukui, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kurume University Hospital, Fukuoka, Kurume
  - Gifu Municipal Hospital, Gifu, Gifu
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - Nagano Municipal Hospital, Hanishina-gun
  - Hiroshima Red Cross Hospital and Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo Kosei General Hospital, Hokkaido, Sapporo
  - Japan Community Health Care Organization Hokkaido Hospital, Hokkaido, Sapporo
  - Tokyo Medical University Ibaraki Medical Center, Ibaraki, Inashiki-gun
  - Tokai University Hospital, Isehara
  - Kanazawa University Hospital, Ishikawa, Kanazawa
  - Shimane University Hospital, Izumo
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Shin-yurigaoka General Hospital, Kanagawa, Kawasaki
  - Kagawa University Hospital, Kita-gun
  - Kobe University Hospital, Kobe
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto Shinto General Hospital, Kumamoto, Kumamoto
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Japanese Red Cross Musashino Hospital, Musashino
  - Shinshu University Hospital, Nagano, Matsumoto
  - Nagasaki Medical Center, Nagasaki, Omura
  - Nara Medical University Hospital, Nara, Kashihara
  - Hyogo College of Medicine Hospital, Nishinomiya
  - The University of Osaka Hospital, Osaka, Suita
  - Oita Cardiovascular Hospital, Ōita
  - Saga University Hospital, Saga
  - Osaka Rosai Hospital, Sakai
  - Seichokai Bell Land General Hospital, Sakai
  - Sendai Tokushukai Hospital, Sendai
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Juntendo University Shizuoka Hospital, Shizuoka, Izunokuni
  - Suita Hospital, Suita-Shi
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Juntendo University Hospital, Tokyo
  - Institute of Science Tokyo Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toranomon Hospital, Tokyo, Minato-ku
  - Mie University Hospital, Tsu
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama City University Hospital, Yokohama
- Jordan (2):
  - The Speciality Hospital (TSH), Amman
  - Jordan University Hospital, Jordan
- Kazakhstan (2):
  - Institute of Gastroenterology, Gepatology and Metabolism LLP, Almaty
  - Asfendiyarov Kazakh National Medical University, Almaty
- Malaysia (4):
  - Hospital Ampang, Ampang
  - Hospital Universiti Sains Malaysia, Kota Bharu
  - University of Malaya Medical Centre, Kuala Lumpur
  - Queen Elizabeth Hospital, Putrajaya
- Mexico (6):
  - Centro de Investigacion Clinica del Pacifico (CICPA), Acapulco de Juárez
  - Clinicos Asociados BOCM SC, Benito Juarez, Mexico
  - Centro de Investigación y Gastroenterología, Col. Xoco
  - Centro de Investigación y Gastroenterología, Mexico City
  - Medical Care and Research, Mérida
  - Practice Dr Rosa Isela Luna Ceballos, Veracruz
- New Zealand (4):
  - New Zealand Clinical Research (NZCR), Grafton, Auckland
  - Middlemore Hospital, Papatoetoe, Auckland
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Waikato Region
- Poland (9):
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Santa SP. z o.o, Lodz
  - FutureMeds Lodz, Lodz
  - Uniwersytecki Szpital Kliniczny Nr 1 W Lublinie, Lublin
  - ID Clinic, Mysłowice
  - FutureMeds Warszawa Centrum, Warsaw
  - Bodyclinic sp. z o.o. sp.k., Warsaw
  - FutureMeds Wroclaw, Wroclaw
  - EMC Instytut Medyczny S.A. - Wroclaw, Wroclaw
- Puerto Rico (3):
  - Klinical Investigations Group, LLC, San Juan
  - Latin Clinical Trial Center, San Juan
  - FDI Clinical Research, San Juan
- Romania (2):
  - Regional Institute of Gastroenterology Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca
  - Spital Judetean De Urgenta Satu Mare, Satu Mare
- Saudi Arabia (2):
  - King Faisal Specialist Hospital and Research Center, Riyadh
  - King Abdulaziz Medical City, National Guard Health Affairs, Riyadh
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Africa (2):
  - Practice Dr Naeem Moosa, Johannesburg
  - Inspired GI Care, Plumstead
- South Korea (10):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Pusan National University Hospital, Busan
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Clínico de Santiago, Santiago de Compostela
- Switzerland (3):
  - Fondazione Epatocentro Ticino, Arzo
  - Hopitaux Universitaires de Geneve (HUG), Geneva
  - University Hospital Zurich, Zurich
- Taiwan (10):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsuing City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation (CGMF) - Linkou Bran, Taoyuan
- Turkey (Türkiye) (8):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Fatih
  - Koc Universitesi Hastanesi, Istanbul
  - Memorial Bahçelievler Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Recep Tayyip Erdogan Universitesi Egitim ve Arastirma Hastanesi, Rize
- United Kingdom (25):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Velocity Clinical Research, Bristol, Bristol
  - Elpida Clinical Trials - Parsloes Hub, Dagenham
  - Derby City General Hospital, Derby
  - Elpida Clinical Trials - Edgware Community Hospital, Edgware
  - Royal Devon and Exeter Hospital, Wonford, Exeter
  - Frimley Park Hospital NHS Foundation Trust, Frimley
  - Panthera Biopartners - Glasgow, Glasgow
  - St Luke's Cancer Centre, Guildford
  - Aintree University Hospital, Liverpool
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Chelsea and Westminster Hospital NHS Foundation Trust - Chelsea and Westminster Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Accellacare North London, Northwood
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Accellacare - Orpington, Orpington
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Manchester, Rochdale
  - Panthera Biopartners - Sheffield, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Elpida Sciences Clinical Trials, Wigan
  - Panthera Biopartners - York, York

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com